CLINICAL TRIAL: NCT03413345
Title: Effect of Rehabilitation on Ejection Fraction (FE) in Cardiopathic and Non Cardiopathic Patients Undergoing Major Orthopedic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Epiq7CC2013
Record Dates: First submitted 2017-12-19; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects without a history of cardiac disease
- subjects with a history of cardiac disease

SUMMARY:
It is a trial aimed to evaluate the ejection fraction in the preoperative phase and during follow-up in two groups of subjects undergoing major orthopedic surgery: the first consisting of subjects without history of cardiac disease, and the second from subjects with a history of cardiopulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* Age: < or equal 18 and > or equal 85 years
* major orthopedic surgery
* rehabilitation at our site
* a positive history for the cardiopathic group

Exclusion Criteria:

* Age: > 85 and < 18
* impossibility to participate to the rehabilitative protocol or come to the follow up visit
* lack of consensus
* previous acute cerebrovascular and / or cardiological events within 6 months prior to enrollment
* previous myocardial (percutaneous and / or surgical) revascularization interventions within the 6 months prior to enrollment
* previous (even in pediatric age) interventions of surgical correction of congenital heart disease
* severe heart failure
* reimplantation of prosthesis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the population consists of 188 subjects (94 subjects for the cardiopathic arm and 94 subjects for the non-cardiopathic arm) undergoing to major orthopedic surgery (hip and knee prosthesis)
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-09-23 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2019-01-18 (Estimated)

PRIMARY OUTCOMES:
Effect of rehabilitation on the ejection fraction (FE) in cardiopathic and non-cardiac patients undergoing major orthopedic surgery | 6 months
  Left ventricular evaluation of ejection fraction (FE) at 6 months in cardiopathic patients with vitamin D deficiency subjected to supplementation with calcifediol

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy